CLINICAL TRIAL: NCT00069888
Title: A Multicenter, Open-Label, Phase II Trial of Adjuvant Taxotere in Patients At High Risk of Relapse Following Prostatectomy
Brief Title: A Phase II Trial of Adjuvant Docetaxel in Patients At High Risk of Relapse Following Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976J_2501; NCT00054509 (obsolete NCT alias)
Record Dates: First submitted 2003-10-02; First posted 2003-10-06 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: Docetaxel

SUMMARY:
This clinical trial is designed to study whether docetaxel (Taxotere) helps reduce the risk of relapse in patients with prostate cancer who have had their prostate removed by surgery, but are at high risk of their cancer recurring. During the trial, doctors will also closely monitor patients for side effects of the chemotherapy.

Docetaxel is a chemotherapy drug that prevents tumor cells from dividing, so they stop growing or die. Doctors use docetaxel to treat lung and breast cancer, and studies show it can help shrink tumors in some patients with prostate cancer that has spread to other parts of their bodies. The researchers conducting this study want to determine if docetaxel also helps reduce the likelihood of prostate cancer returning after surgery has removed the original tumor.

All of the study participants will receive up to 18 doses of docetaxel, each administered through a needle inserted into a vein. Each round of treatment will consist of 30-minute, weekly infusions for three consecutive weeks, followed by one week with no chemotherapy. Before and after the chemotherapy, patients will take dexamethasone, an oral steroid that reduces the risk of an allergic reaction to the medication. If the side effects of the treatment become too intense, doctors may modify, delay, or even stop chemotherapy during the trial.

ELIGIBILITY:
INCLUSION CRITERIA:

* patients with prostate cancer who have just undergone prostatectomy,
* high risk of their cancer recurring (High risk is defined as at least a 50 percent chance the cancer will return within three years after surgery.)

EXCLUSION CRITERIA:

* Prior systemic treatment for prostate cancer with hormonal therapy, chemotherapy, or any other anticancer therapy.
* Prior radiation therapy
* Patients receiving any concurrent therapy for cancer. This includes alternative therapies
* Patients requiring concurrent treatment with corticosteroids, with the exception of inhaled and topical corticosteroids.
* History of a malignancy other than prostate cancer
* Peripheral neuropathy >/= Grade 2
* Psychological, familial, sociological or geographical conditions which do not permit treatment and/or medical follow-up required to comply with the study protocol
* Patients with a history of hypersensitivity reaction to products containing Polysorbate 80 (Tween 80).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2001-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To assess the preliminary effects of six cycles of adjuvant, weekly Taxotere® (three weeks on/one week off) on the rate of progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Nagarwala, M.D., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis US, Bridgewater, New Jersey, United States